CLINICAL TRIAL: NCT03395457
Title: A Pragmatic Randomised Controlled Trial on the Effectiveness of Manual Therapy as an Adjunct to Tertiary Management in Chronic Migraine
Brief Title: Tertiary Care With or Without Manual Therapy for Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bournemouth 228901
Record Dates: First submitted 2018-01-03; First posted 2018-01-10 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Chronic Migraine
MeSH Terms: interventions — Dosage Forms; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: pragmatic randomised control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care as usual (Active Comparator): This is the care provided by the neurologist for chronic migraine.
  Interventions: Drug: Care as usual
- Care as usual plus manual therapy (Experimental): Other
  Interventions: Drug: Care as usual; Other: Manual Therapy

INTERVENTIONS:
Drug: Care as usual — Application of usual pharmacological care for chronic migraine
  Other Names: Medication for chronic migraine
Other: Manual Therapy — 5 sessions of manual therapy over 12 weeks
  Arms: Care as usual plus manual therapy

SUMMARY:
The aim of this study is to determine if adding manual therapy to care as usual reduces the discomfort from chronic migraine compared to care as usual alone

ELIGIBILITY:
Inclusion Criteria:

Female adults 18 years of age or older with a good command of English (to enable informed consent) Existing patients with chronic migraine as diagnosed by a clinical interview with a neurologist in line with the International Classification of Headache Diagnosis criteria (ICHD) Undergoing care as usual from the neurologist

Exclusion Criteria:

Currently having or had manual therapy for neck, shoulder in the last six weeks.

Having a condition contraindicated for manual therapy including but not limited to inflammatory disorders, severe osteoporosis and tumours.

Identification of any medical 'red flags' by the neurologist including

* Evidence of any central nervous system involvement for example:
* Facial palsy (presence of ptosis/Horner's syndrome)
* Visual disturbance (presence of blurred vision, diplopia, hemianopia)
* Speech disturbance (presence of dysarthria, dysphonia, dysphasia such as expressive or receptive)
* Balance disturbance (presence of dizziness, imbalance, unsteadiness, falls)
* Paraesthesia (presence, location such as upper limb/lower limb, face)
* Weakness (presence, location such as upper limb/lower limb)
* Known major psychiatric or psychological conditions not under control

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in migraine-related disability | 12 weeks
  Headache Impact Test (HIT6). The six-item Headache Impact Test (HIT-6) provides a global measure of adverse headache impact and is used in screening and monitoring patients. The HIT-6 items measure the adverse impact of headache on social functioning, role functioning, vitality, cognitive functioning, psychological distress and the severity of headache pain.
  The final HIT-6 score is obtained from simple summation of the six items and ranges between 36 and 78, with larger scores reflecting greater impact. The categories used for interpretation of impact are: little or no impact (49 or less), some impact (50-55), substantial impact (56-59), and severe impact (60-78).

SECONDARY OUTCOMES:
Change in Migraine Specific Quality of Life Questionnaire Score (MSQoL 2.1) | 12 weeks
  The 14-item instrument measures how migraines affect daily functioning across three domains: Role function Restrictions (7 items assessing how migraines limit one's daily social and work-related activities); Role function prevention (4 items assessing how migraines prevent these activities); Emotional Functional (3 items assessing the emotions associated with migraines). It uses a 6-point scale: "none of the time," "a little bit of the time," "some of the time," "a good bit of the time," "most of the time," and "all of the time," which are assigned scores of 1 to 6, respectively. Scores are computed as a sum of item responses and rescaled from a 0 to 100 scale such that higher scores indicate better quality of life.
Headache Frequency | 12 weeks
  Percentage of participants with reduction in headache frequency of greater than 50%

CONTACTS AND LOCATIONS:
Overall Officials: Carol Clark, Dr, Study Chair — University Bournemouth
Locations (1):
- Salford Royal NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] Odell J, Clark C, Hunnisett A, Ahmed OH, Branney J. Manual therapy for chronic migraine: a pragmatic randomised controlled trial study protocol. Chiropr Man Therap. 2019 Mar 27;27:11. doi: 10.1186/s12998-019-0232-4. eCollection 2019. PMID 30962877